CLINICAL TRIAL: NCT03551158
Title: The Search for Non-invasive Determinants of Response to Ablation of Atrial Fibrillation. Non-invasive Evaluation of Left Atrium Anatomy and Function With Three Dimensional Echocardiography: Comparison With Cardiac CT and MRI
Brief Title: Non - Invasive Evaluation of the Left Atrium Anatomy and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017/221
Record Dates: First submitted 2018-02-27; First posted 2018-06-11 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2017-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atrial fibrillation patients (Other): Patients with atrial fibrillation who underwent cryoballoon ablation
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Cardiac imaging for the assessment of the left atrium anatomy and function.
  Other Names: cardiac computed tomography; cardiac magnetic resonance

SUMMARY:
The aim of the study is to evaluate the accuracy and reproducibility of the left atrium (LA) anatomy and function in different populations and in patients with atrial fibrillation who have undergone cryoballoon ablation.

DETAILED DESCRIPTION:
This study implies three parts. The first part of the study aims to evaluate the variability and reproducibility of rest two - and three-dimensional echocardiography for the left atrium anatomy and function and to assess their correlation with clinical variables.

The second part of the study aims to evaluate the accuracy and reproducibility of the left atrium anatomy and function using echocardiography and to validate it with cardiac CT. Moreover, the study aims to evaluate which parameters can predict the recurrence of atrial fibrillation in patients who have undergone atrial fibrillation ablation.

The third part of the study aims to assess the accuracy and variability of echocardiographic measurements compared to cardiac magnetic resonance and to find predictors of recurrence after cryoballoon ablation for atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* subsequent group of patients sent to the echocardiography laboratory for any indication/patients who have undergone a cryoballoon ablation
* older than 18 years old

Exclusion Criteria:

• inadequate image quality during echocardiography, contraindications for computed tomography or cardiac magnetic resonance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence | 1 year
  Predictors of atrial fibrillation recurrence after ablation

CONTACTS AND LOCATIONS:
Overall Officials: Steven Droogmans, Professor, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoit BD. Left atrial size and function: role in prognosis. J Am Coll Cardiol. 2014 Feb 18;63(6):493-505. doi: 10.1016/j.jacc.2013.10.055. Epub 2013 Nov 27. PMID 24291276
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Garg J, Chaudhary R, Palaniswamy C, Shah N, Krishnamoorthy P, Bozorgnia B, Natale A. Cryoballoon versus Radiofrequency Ablation for Atrial Fibrillation: A Meta-analysis of 16 Clinical Trials. J Atr Fibrillation. 2016 Oct 31;9(3):1429. doi: 10.4022/jafib.1429. eCollection 2016 Oct-Nov. PMID 28496925
- [Background] Gerede DM, Candemir B, Vurgun VK, Aghdam SM, Acibuca A, Ozcan OU, Goksuluk H, Kervancioglu C, Erol C. Prediction of recurrence after cryoballoon ablation therapy in patients with paroxysmal atrial fibrillation. Anatol J Cardiol. 2015 Sep 15;16(7):482-8. doi: 10.5152/AnatolJCardiol.2015.6309. Online ahead of print. PMID 26680545
- [Background] Badano LP, Pezzutto N, Marinigh R, Cinello M, Nucifora G, Pavoni D, Gianfagna P, Fioretti PM. How many patients would be misclassified using M-mode and two-dimensional estimates of left atrial size instead of left atrial volume? A three-dimensional echocardiographic study. J Cardiovasc Med (Hagerstown). 2008 May;9(5):476-84. doi: 10.2459/JCM.0b013e3282f194f0. PMID 18403999
- [Background] Nedios S, Kosiuk J, Koutalas E, Kornej J, Sommer P, Arya A, Richter S, Rolf S, Husser D, Hindricks G, Bollmann A. Comparison of left atrial dimensions in CT and echocardiography as predictors of long-term success after catheter ablation of atrial fibrillation. J Interv Card Electrophysiol. 2015 Sep;43(3):237-44. doi: 10.1007/s10840-015-0010-8. Epub 2015 May 9. PMID 25956477
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2015 Mar;16(3):233-70. doi: 10.1093/ehjci/jev014. PMID 25712077
- [Background] Badano LP, Miglioranza MH, Mihaila S, Peluso D, Xhaxho J, Marra MP, Cucchini U, Soriani N, Iliceto S, Muraru D. Left Atrial Volumes and Function by Three-Dimensional Echocardiography: Reference Values, Accuracy, Reproducibility, and Comparison With Two-Dimensional Echocardiographic Measurements. Circ Cardiovasc Imaging. 2016 Jul;9(7):e004229. doi: 10.1161/CIRCIMAGING.115.004229. PMID 27412658
- [Background] Mor-Avi V, Yodwut C, Jenkins C, Kuhl H, Nesser HJ, Marwick TH, Franke A, Weinert L, Niel J, Steringer-Mascherbauer R, Freed BH, Sugeng L, Lang RM. Real-time 3D echocardiographic quantification of left atrial volume: multicenter study for validation with CMR. JACC Cardiovasc Imaging. 2012 Aug;5(8):769-77. doi: 10.1016/j.jcmg.2012.05.011. PMID 22897989
- [Background] Todaro MC, Choudhuri I, Belohlavek M, Jahangir A, Carerj S, Oreto L, Khandheria BK. New echocardiographic techniques for evaluation of left atrial mechanics. Eur Heart J Cardiovasc Imaging. 2012 Dec;13(12):973-84. doi: 10.1093/ehjci/jes174. Epub 2012 Aug 21. PMID 22909795
- [Background] Agner BF, Kuhl JT, Linde JJ, Kofoed KF, Akeson P, Rasmussen BV, Jensen GB, Dixen U. Assessment of left atrial volume and function in patients with permanent atrial fibrillation: comparison of cardiac magnetic resonance imaging, 320-slice multi-detector computed tomography, and transthoracic echocardiography. Eur Heart J Cardiovasc Imaging. 2014 May;15(5):532-40. doi: 10.1093/ehjci/jet239. Epub 2013 Nov 17. PMID 24247925